CLINICAL TRIAL: NCT04559035
Title: Nasal Irrigation to Reduce COVID-19 Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Matt Lyon, Responsible Party, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1603291
Record Dates: First submitted 2020-09-21; First posted 2020-09-22 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: prevention; nasal lavage; povidone-iodine
MeSH Terms: conditions — COVID-19 | interventions — Nasal Lavage

STUDY DESIGN:
Intervention Model Description: randomized clinical trial of two nasal irrigation protocols in outpatients PCR positive for SARS-CoV-2, nested in a prospective case:cohort using laboratory-confirmed cases in the CDC COVID-19 Case Surveillance dataset
Who Masked: Outcomes Assessor
Masking Description: Hospitalization records were confirmed by study personnel blinded to participant status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betadine (Other): Intervention - twice-a-day nasal lavage Twice-a-day virucidal group: Participants randomized to betadine will receive 2 gallon jugs of distilled water, two NeilMed Sinus Irrigation bottles and 28 salination packets (with some extras), OR one Navage unit with 28 SaltPods (and some extras), and a cardboard receptacle labeled "used saline containers" to keep track of adherence.
  Those randomized to receive betadine will also receive one bottle of povidone-iodine, a one-sheet instruction with photographs demonstrating how to add ½ tsp betadine in addition to the salination packet to the sinus irrigation bottle or Navage unit reservoir prior to SaltPod, along with a ½ tsp measuring spoon.
  Interventions: Other: Nasal lavage
- Baking Soda (Other): Twice-a-day alkalinized group: Participants randomized to alkalinization will receive 2 gallon jugs of distilled water, two Neilmed bottles with 28 saline packets, OR one Navage unit with 28 SaltPods, and a cardboard receptacle labeled "used saline containers" to keep track of adherence. Those randomized to alkalinization will also receive a box of baking soda, ½ tsp measuring spoon and instructions on how to add the baking soda.
  Interventions: Other: Nasal lavage

INTERVENTIONS:
Other: Nasal lavage — Twice daily nasal lavage.

SUMMARY:
The purpose of this study is to evaluate if using nasal irrigation, also known as nasal lavage, for 14 days after a positive test in high risk patients can reduce the severity of symptoms associated with COVID-19. Nasal lavage consists of running salt water in one nostril and out the other to get rid of germs. Nasal irrigation was done with either Betadine or baking soda to determine if adding an antimicrobial or changing the pH of the mucous helped. Hospitalization and death were compared for combined nasal irrigation groups to the CDC dataset of patients aged 50+

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if using nasal irrigation, also known as nasal lavage, can reduce the severity of symptoms associated with COVID-19. Nasal lavage consists of running salt water in one nostril and out the other to get rid of germs. Saline nasal irrigation with Betadine or baking soda will be evaluated.

Participants will be asked to do several things during this study: watch a one minute video on YouTube, use a nasal irrigation device twice a day for 14 days, complete a one-time detailed survey and keep a research diary about their usage and symptoms using an on-line application called Qualtrics, agree to be texted reminders, be called on the phone if they fail to complete the daily diary two days in a row, agree to be called four times, and provide contact information for a secondary person who can be contacted if the primary participant is unavailable.

Participation in this study does not involve any significant risks. However, some people may find using nasal irrigation causes them some discomfort.

While there are no known benefits to participating in the study participants may see a reduction in their symptoms more quickly than if they didn't participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and providing informed consent using remote consent
* Willingness and physical capacity to initiate nasal irrigation and to adhere to the protocol
* Willing to give additional contact phone number of another person who will know the health status of the participant and agree to be contacted if needed for follow-up
* 55 years of age or older
* Has access to and the willingness and ability to adhere to the technological requirement of the study i.e. able to use a smartphone for voice and text and email and access to the internet at home
* English speaking
* Positive rapid COVID-19 test performed the day of or the day before enrollment

Exclusion Criteria:

* Currently doing daily nasal irrigation
* Current supplemental oxygen therapy
* Unwillingness to try nasal irrigation or use nasal irrigation twice a day
* Nasal surgery within the past year or chronic sinusitis
* Prior COVID-19 infection or positive test >1 day before present
* Symptoms longer than 7 days prior to testing as reported to researchers
* Allergy to iodine or shellfish
* Participation in another prospective COVID related research project (clinical trial).
* Employed and working as a healthcare worker.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Frequency | 28 days
  Rate of hospitalization by number of episodes of nasal irrigation out of 28 possible.
  To assess reduction in admission, in patients with differing nasal irrigation frequency over 14 days with an additional 14 day follow-up period.

SECONDARY OUTCOMES:
Reduction | 28 days
  Reduction of severity of COVID outcomes by number of episodes of nasal irrigation out of 28 possible.
  Assess reduction in hospital visits, symptoms, supplemental oxygen use, ICU admission, and death in patients with differing nasal irrigation frequency.
  Reduction of severity of COVID outcomes by nasal irrigation with alkalination or virucidal additives.
  To assess reduction in admission, hospital visits, symptoms, supplemental oxygen use, ICU admission, and death in patients using alkalnization or virucidal additives to nasal irrigation over 14 days with an additional 14 day follow-up period, controlling for irrigation frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Lyon, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frank S, Capriotti J, Brown SM, Tessema B. Povidone-Iodine Use in Sinonasal and Oral Cavities: A Review of Safety in the COVID-19 Era. Ear Nose Throat J. 2020 Nov;99(9):586-593. doi: 10.1177/0145561320932318. Epub 2020 Jun 10. PMID 32520599
- [Background] Pelletier JS, Tessema B, Frank S, Westover JB, Brown SM, Capriotti JA. Efficacy of Povidone-Iodine Nasal and Oral Antiseptic Preparations Against Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV-2). Ear Nose Throat J. 2021 Apr;100(2_suppl):192S-196S. doi: 10.1177/0145561320957237. Epub 2020 Sep 21. PMID 32951446
- [Background] Bidra AS, Pelletier JS, Westover JB, Frank S, Brown SM, Tessema B. Rapid In-Vitro Inactivation of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Using Povidone-Iodine Oral Antiseptic Rinse. J Prosthodont. 2020 Jul;29(6):529-533. doi: 10.1111/jopr.13209. Epub 2020 Jun 16. PMID 32511851
- [Background] Frank S, Brown SM, Capriotti JA, Westover JB, Pelletier JS, Tessema B. In Vitro Efficacy of a Povidone-Iodine Nasal Antiseptic for Rapid Inactivation of SARS-CoV-2. JAMA Otolaryngol Head Neck Surg. 2020 Nov 1;146(11):1054-1058. doi: 10.1001/jamaoto.2020.3053. PMID 32940656
- [Background] Seet RCS, Quek AML, Ooi DSQ, Sengupta S, Lakshminarasappa SR, Koo CY, So JBY, Goh BC, Loh KS, Fisher D, Teoh HL, Sun J, Cook AR, Tambyah PA, Hartman M. Positive impact of oral hydroxychloroquine and povidone-iodine throat spray for COVID-19 prophylaxis: An open-label randomized trial. Int J Infect Dis. 2021 May;106:314-322. doi: 10.1016/j.ijid.2021.04.035. Epub 2021 Apr 20. PMID 33864917
- [Background] Anderson DE, Sivalingam V, Kang AEZ, Ananthanarayanan A, Arumugam H, Jenkins TM, Hadjiat Y, Eggers M. Povidone-Iodine Demonstrates Rapid In Vitro Virucidal Activity Against SARS-CoV-2, The Virus Causing COVID-19 Disease. Infect Dis Ther. 2020 Sep;9(3):669-675. doi: 10.1007/s40121-020-00316-3. Epub 2020 Jul 8. PMID 32643111
- [Background] Guenezan J, Garcia M, Strasters D, Jousselin C, Leveque N, Frasca D, Mimoz O. Povidone Iodine Mouthwash, Gargle, and Nasal Spray to Reduce Nasopharyngeal Viral Load in Patients With COVID-19: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Apr 1;147(4):400-401. doi: 10.1001/jamaoto.2020.5490. PMID 33538761
- [Background] Singh A, Yadav M, Sikka K. Regarding Use of Povidone Iodine to Reduce Nasopharyngeal Viral Load in Patients With COVID-19. JAMA Otolaryngol Head Neck Surg. 2021 Jul 1;147(7):680-681. doi: 10.1001/jamaoto.2021.0683. No abstract available. PMID 33914069

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT04559035/Prot_SAP_ICF_000.pdf